CLINICAL TRIAL: NCT05780554
Title: Post-transplantation Cyclophosphamide in Haploidentical Stem Cell Allografts Dose Reduction: 50 mg/kg vs 25 mg/kg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Centro de Hematología y Medicina Interna (Other)
Responsible Party: Principal Investigator, Guillermo J. RUIZ-ARGÜELLES, General director, Centro de Hematología y Medicina Interna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHMI-020323-1
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Graft Vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclophosphamide 50 mg/kg (Active Comparator)
  Interventions: Drug: Cyclophosphamide
- Cyclophosphamide 25 mg/kg (Experimental)
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — Post transplant cyclophosphamide 25 mg/kg on day +3 and +4
  Arms: Cyclophosphamide 25 mg/kg
Drug: Cyclophosphamide — Post transplant cyclophosphamide 50 mg/kg on day +3 and +4
  Arms: Cyclophosphamide 50 mg/kg

SUMMARY:
Allogeneic hematopoietic cell transplantation (HSCT) is a worldwide recognized therapy for several hematologic malignancies; a modality extensively used around the world due to its effectivity; however, an HLA-matched sibling or unrelated donor is not always available, because of diverse factors such as: ethnic minorities and multiethnic families, socio-economic status, among others. This problem has led to an expansion of the donor pool to include alternative donor sources such as HLA-haploidentical (Haplo) relatives, HLA-mismatched unrelated donors, and HLA-matched or mismatched cord blood.

In the Hematology and Internal Medicine Center of Clinica Ruiz, we have seen that 50% reduced doses of post-transplantation cyclophosphamide (25 mg/Kg) on days +3 and +4 have a favorable effect on patient's survival rates compared to the full 50 mg/Kg doses. Haplo-HSCT can be conducted safely on an outpatient basis, using peripheral blood stem cells, this leading into substantial decreases in the costs. Outpatient-based Haplo-HSCT has turned into the solution of the HSCT most frequent problems in low- and middle-income countries (LMIC): Cost and donor availability. The high dose administration of PT-Cy after transplant can lead into hematological and cardiac, toxicities. There is preliminary information about diminished doses of PTCy, might being equally effective in the prevention of GVHD and substantially less toxic.

ELIGIBILITY:
Inclusion Criteria:

* Candidates to receive a Haplo-HSCT (myeloid acute leukemia, lymphoid acute leukemia, myelodysplastic syndrome, multiple myeloma, Hodgkin lymphoma, non-Hodgkin lymphoma, myeloid chronic leukemia, medullary hypoplasia, non-malignant hematologic diseases).
* Patients able to travel to and remain in Puebla, México during a 4-week period, accompanied by a caregiver.

Exclusion Criteria:

* Patients who refuse to sign the consent form.
* Latent infection.
* Hepatic, cardiac or bronchopulmonary symptomatic diseases
* Abnormalities on previous clinical hematological appointments, considered as contraindication.
* Positive serology for HIV, VHB, VHC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Acute GVHD rate | 6 months
  Incidence of acute GVHD after HSCT
Chronic GVHD rate | 18 months
  Incidence of chronic GVHD after HSCT
Relapse free survival | 12 months
  Incidence of relapse of the disease after HSCT
Overall survival | 12 months
  Patients survival after therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Hematología y Medicina Interna, Puebla City, Mexico

REFERENCES:
- [Derived] Olivares-Gazca JC, Pastelin-Martinez ML, Montes-Robles MA, Gallardo-Perez MM, Hernandez-Flores EJ, Robles-Nasta M, Sanchez-Bonilla D, Ruiz-Delgado GJ, Ruiz-Arguelles GJ. Can doses of post-transplantation cyclophosphamide in haploidentical stem cell allografts be reduced? Hematology. 2023 Dec;28(1):2242176. doi: 10.1080/16078454.2023.2242176. PMID 37530697